CLINICAL TRIAL: NCT06409247
Title: Testing the Role of Attentional and Audio Vocal Mechanisms in a New Internet- Based Intervention for Social Anxiety: iExposure
Brief Title: iExposure Intervention for Social Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto University (Other)
Responsible Party: Principal Investigator, Mikael Rubin, Assistant Professor, Palo Alto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-052-PAU
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Social Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard iExposure (Active Comparator): iExposure. Participants will complete four intervention sessions within two weeks. The intervention will use an entirely self-guided protocol delivered via Qualtrics and Gorilla Experiment Builder:
  1. During the first session, participants will receive a brief standardized psychoeducation module, presented via a 15-minute video recording. This video will explain the intervention, its rationale, and the procedure.
  2. Participants will then complete 10 simulated teleconferencing interaction trials with different topics, each lasting a maximum of two minutes. During each call participants will be prompted by one of the audience members to respond to a question (described in further detail in the Materials section, below).
  3. Participants will complete the Subjective Units of Distress Scale before and after each speech trial.
  4. Sessions 2-4 involve the same protocol and the four intervention sessions are completed within two weeks.
  Interventions: Behavioral: iExposure
- iExposure + Attention Guidance Augmentation (Experimental): Attention Guidance Augmentation. The attention guidance condition consists of two unique components in addition to the standard iExposure intervention: (1) the intervention rationale will include information about the importance of visually attending to the faces of the audience; (2) participants will be given a target audience member to focus their gaze on during each impromptu response. They will be told that they should look at and focus on the target audience member for the whole response. In each progressive session the number of trials where the participant is directed to focus on an uninterested audience member will increase.
  Interventions: Behavioral: iExposure plus attention guidance
- iExposure + Attention Control Augmentation (Experimental): The attention control condition consists of two unique components in addition to the standard iExposure intervention (1) the intervention rationale will include information about the importance of developing attention control; (2) participants will be given a central region of the screen (non-audience member) to focus on. They will be told that they should look at and focus on the central region for the whole response.
  Interventions: Behavioral: iExposure plus attention control

INTERVENTIONS:
Behavioral: iExposure — There will be 4 treatment sessions, covering the iExposure intervention. The intervention and assessment process is entirely self-guided. Each session will last approximately 60 minutes. Participants will complete 10 mock-interaction trials for each session.
  Arms: Standard iExposure
Behavioral: iExposure plus attention guidance — The attention guidance condition consists of two unique components in addition to the standard iExposure intervention: (1) the intervention rationale will include information about the importance of visually attending to the faces of the audience; (2) participants will be given a target audience member to focus their gaze on during each impromptu response. They will be told that they should look at and focus on the target audience member for the whole response. In each progressive session the number of trials where the participant is directed to focus on an uninterested audience member will increase.
  Arms: iExposure + Attention Guidance Augmentation
Behavioral: iExposure plus attention control — The attention control condition consists of two unique components in addition to the standard iExposure intervention (1) the intervention rationale will include information about the importance of developing attention control; (2) participants will be given a central region of the screen (non-audience member) to focus on. They will be told that they should look at and focus on the central region for the whole response.
  Arms: iExposure + Attention Control Augmentation

SUMMARY:
Social anxiety (SA) is a highly prevalent mental health concern, thought to disproportionately affect youth with recent international estimates of more than 30% of individuals reporting clinically elevated symptoms. Despite the prevalence of SA, as few as one in five individuals receive care, due to limited access to evidence-based treatments. Additionally there has been a notable increase in social anxiety since the start of the COVID-19 pandemic. This proposal will use iExposure to develop a personalized mechanism-focused approach to optimizing treatment response for individuals with social anxiety by testing standard iExposure against two augmentations that incorporate distinct attention mechanisms (attention guidance and attention control).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Fluent in English
* Leibowitz Social Anxiety Scale > 47 and endorses both social anxiety items on the Web Screening Questionnaire for Common Mental Disorders

Exclusion Criteria:

* Currently receiving CBT for Social Anxiety Disorder
* Significant visual impairment precluding engagement in the simulated teleconferencing interactions
* Unstable dose of psychotropic medications within 6 weeks prior to baseline assessment
* Current alcohol or substance use disorder
* Current or past bipolar disorder or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale Self Report Version | 0 days
  The Liebowitz Social Anxiety Scale Self Report Version is a 48-item self-report measure of fear and avoidance concerning social interactions and performance situations (e.g., telephoning in public, talking to people in authority). The range of scores is 0-144; higher scores are worse.
Liebowitz Social Anxiety Scale Self Report Version | 15 days
  The Liebowitz Social Anxiety Scale Self Report Version is a 48-item self-report measure of fear and avoidance concerning social interactions and performance situations (e.g., telephoning in public, talking to people in authority). The range of scores is 0-144; higher scores are worse.
Liebowitz Social Anxiety Scale Self Report Version | 45 days
  The Liebowitz Social Anxiety Scale Self Report Version is a 48-item self-report measure of fear and avoidance concerning social interactions and performance situations (e.g., telephoning in public, talking to people in authority). The range of scores is 0-144; higher scores are worse.
Personal Report of Communication Apprehension (PRCA) | 0 days
  The Personal Report of Communication Apprehension is a 24-item that assesses anxiety related to speaking in a variety of situation. The range of scores is 24-120; higher scores are worse.
Personal Report of Communication Apprehension | 15 days
  The Personal Report of Communication Apprehension is a 24-item that assesses anxiety related to speaking in a variety of situation. The range of scores is 24-120; higher scores are worse.
Personal Report of Communication Apprehension | 45 days
  The Personal Report of Communication Apprehension is a 24-item that assesses anxiety related to speaking in a variety of situation. The range of scores is 24-120; higher scores are worse.

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale - Revised | 0 days
  The Center for Epidemiologic Studies Depression Scale - Revised is a 20-item measure of depression. The range of scores is 0-60; higher scores are worse.
Center for Epidemiologic Studies Depression Scale - Revised | 15 days
  The Center for Epidemiologic Studies Depression Scale - Revised is a 20-item measure of depression. The range of scores is 0-60; higher scores are worse.
Center for Epidemiologic Studies Depression Scale - Revised | 45 days
  The Center for Epidemiologic Studies Depression Scale - Revised is a 20-item measure of depression. The range of scores is 0-60; higher scores are worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared as part of the National Institute of Mental Health Data Archive
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: All publications will be posted to the PubMed database, consistent with the National Institutes of Health Public Access Policy and have an NDA study linking the analytical output to the underlying data collection, including a description of the analytic methodology, derived variables, and the statistical/analytical model outputs. Each of these studies is assigned a digital object identifier (DOI). This data DOI will be included in any resulting manuscripts to facilitate easy access to the data used for the publication. Data not previously shared through an NDA study will be made available at the end of the project period. Researchers will request data using standard NDA application processes, and the NDA committee will decide which requests are provided. The standard NDA access process allows access for one year and is renewable. Once the data are submitted to NDA, NDA will control the long-term persistence of the data.
Access Criteria: Access will be controlled by the National Institute of Mental Health Data Archive Data Access Committee